CLINICAL TRIAL: NCT06974656
Title: Intraoperative Intravenous Infusion of Dexmedetomidine Versus Lidocaine in Management of Acute Postoperative Pain After Modified Radical Mastectomy: A Randomized Trial
Brief Title: Infusion of Dexmedetomidine Versus Lidocaine in Management of Acute Postoperative Pain After Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Elsaid Abdel Fattah, Lecturer of Anesthesia, Surgical ICU and Pain Management, Faculty of Medicine, National Cancer Institute, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2503-501-100-197
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Infusion; Dexmedetomidine; Lidocaine; Acute; Postoperative Pain; Modified Radical Mastectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Patients will receive 1 μg/kg of intravenous dexmedetomidine over 10 min followed by an intravenous infusion of n 0.3-0.5 μg/kg/h.
  Interventions: Drug: Dexmedetomidine
- Lidocaine group (Experimental): Patients will receive a bolus of intravenous lidocaine 1.5mg/kg over 10 min followed by a continuous infusion of lidocaine 1.5-2 mg/kg/h.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive 1 μg/kg of intravenous dexmedetomidine over 10 min followed by an intravenous infusion of n 0.3-0.5 μg/kg/h.
  Arms: Dexmedetomidine group
Drug: Lidocaine — Patients will receive a bolus of intravenous lidocaine 1.5mg/kg over 10 min followed by a continuous infusion of lidocaine 1.5-2 mg/kg/h.
  Arms: Lidocaine group

SUMMARY:
This study aims to compare the effect of intraoperative intravenous infusion of dexmedetomidine and lidocaine in the management of acute postoperative pain after mastectomy.

DETAILED DESCRIPTION:
Postoperative pain control continues to remain suboptimal, despite multimodal analgesia regimes, minimally invasive surgical techniques, and enhanced recovery programs. Acute postoperative pain hinders patients' functional recovery and represents one of the greatest predictive factors for transition to chronic postsurgical pain.

Among adjuvants, dexmedetomidine, a highly selective α2 adrenoreceptor agonist, and lidocaine, a well-established local anesthetic, seem promising for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* American Society of Anesthesiology (ASA) physical status II.
* Body mass index (BMI) 18.5-35 kg/m2.
* Scheduled for modified radical mastectomy.

Exclusion Criteria:

* Patient's refusal.
* Contraindication to the use of local anesthetics.
* Cardiovascular disease.
* Significant renal/hepatic impairment
* Insulin-dependent diabetes mellitus.
* Central nervous system or psychiatric disease.
* Use of opioids/steroids/clonidine/other α2 agonist/analgesics or any drugs acting on the central nervous system during the previous 2 weeks.
* Drug/alcohol abuse.
* Inability to comprehend the pain assessment scale.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Wmone scheduled for modified radical mastectomy
Enrollment: 40 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 48 hours postoperatively
  Time to the 1st rescue analgesia will be recorded from the end of surgery till first dose of morphine administrated.

SECONDARY OUTCOMES:
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded before infusion (Baseline value), 5,10, 15, 30, 45, and 60 minutes after the operation, and at the end of the operation.
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded before infusion (Baseline value), 5,10, 15, 30, 45, and 60 minutes after the operation, and at the end of the operation.
Total morphine consumption | 48 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the Visual Analogue Scale (VAS)> 3 to be repeated after 30 min if pain persists until the VAS < 4.
Degree of pain | 48 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at post-anesthesia care unit (PACU), 2, 4, 8, 12, 24, 36, and 48 h postoperatively.
Incidence of adverse events | 48 hours postoperatively
  Incidence of adverse events such as hypotension, bradycardia, nausea, vomiting, or any other complications will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.